CLINICAL TRIAL: NCT00064623
Title: A Randomized, Double-Blind, Controlled Dose Finding Study of NGX-4010 for the Treatment of Painful HIV-Associated Distal Symmetrical Polyneuropathy
Brief Title: Study of NGX-4010 for the Treatment of Painful HIV-Associated Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NeurogesX (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C107
Record Dates: First submitted 2003-07-10; First posted 2003-07-11 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-03

CONDITIONS: HIV Infections; Peripheral Nervous System Diseases; Pain
Keywords: Dermal assessment; Pain measurement; Diary; Analgesics/*therapeutic use; Capsaicin/*administration & dosage/adverse effects; HIV Infections/*complications/*drug therapy; Peripheral Nervous System Diseases/*complications/diagnosis/*therapy; Peripheral Nervous System Diseases/drug therapy/*etiology/physiopathology
MeSH Terms: conditions — HIV Infections; Peripheral Nervous System Diseases; Pain

INTERVENTIONS:
Drug: Capsaicin Dermal Patch

SUMMARY:
The purpose of the study is to determine if an investigational drug, NGX-4010 (high-concentration capsaicin patch), is effective in treating painful HIV-associated neuropathy.

DETAILED DESCRIPTION:
The C107 study is a randomized, double-blind, controlled dose finding study of NGX-4010 for the treatment of painful symptoms of HIV-associated neuropathy. Participants will be randomly assigned to receive initial treatment according to one of three doses (application durations), and to receive double-blind NGX-4010 patch (high-concentration capsaicin) or matching control (low-concentration capsaicin).

Participants who complete study evaluations through Week 12 will have the option of receiving up to 3 additional open-label treatments.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Documented evidence of HIV-1 infection
* Documented diagnosis of painful HIV-associated distal symmetrical polyneuropathy established by a neurologist resulting from HIV disease and/or antiretroviral drug exposure, with primary symptoms of pain, burning or dysesthetic discomfort in both feet for at least 2 months prior to Screening Visit, and absent or diminished ankle reflexes, and at least one of the following: distal diminution of vibration sensation or pain or temperature sensation in the legs
* Either no neurotoxic antiretroviral (didanosine, zalcitabine or stavudine) exposure for at least 8 weeks prior to Screening Visit, or currently on stable dose(s) of any neurotoxic antiretroviral(s) for at least 8 weeks prior to Screening Visit
* Screening Pain Sum Score of 12 to 36
* Karnofsky Performance Score of greater than or equal to 60
* Intact, unbroken skin over the painful area(s) to be treated
* If taking chronic pain medications, be on a stable (not PRN) regimen for at least 21 days prior to Treatment Visit and willing to maintain these medications at the same stable dose(s) and schedule throughout the study
* Female subjects with child-bearing potential: negative serum pregnancy test performed at Screening Visit
* Willing to use effective methods of birth control and/or refrain from participating in a conception process during study and for 30 days following experimental drug exposure
* Willing and able to comply with protocol requirements for duration of study

Exclusion Criteria:

* Concomitant opioid medication, unless orally or transdermally administered and not exceeding a total daily dose of morphine 60 mg/day, or equivalent. Parenteral opioid use is excluded, regardless of dose
* Unavailability of an effective rescue medication strategy for the subject, such as unwillingness to use opioid analgesics during treatment, or high tolerance to opioids precluding the ability to relieve treatment-associated discomfort with Roxicodone® or Vicodin®, as judged by the Investigator
* Active substance abuse or history of chronic substance abuse within the past year, or prior chronic substance abuse judged likely to recur during the study period by the investigator
* Recent use (within 21 days preceding the Treatment Visit of any topically applied pain medication, such as non-steroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics (including Lidoderm®), steroids or capsaicin products on the painful areas
* Current use of any investigational agent or Class 1 anti-arrhythmic drugs
* Significant pain of an etiology other than painful HIV-associated neuropathy; significant ongoing pain from other cause(s) that may interfere with judging HIV-associated neuropathy pain
* Evidence of another contributing cause for peripheral neuropathy, e.g., diabetes mellitus requiring medication control (i.e., oral hypoglycemics, insulin); hereditary neuropathy; vitamin B12 deficiency (B12 level ≤ 200 pg/mL) or less than 3 months of B12 supplementation prior to Screening Visit; or treatment within 90 days prior to Screening Visit with any drug that may have contributed to the sensory neuropathy
* Any implanted medical device (spinal cord stimulator, intrathecal pump or peripheral nerve stimulator) for the treatment of neuropathic pain
* Treatment for acute opportunistic infections within 14 days before Treatment Visit
* Presence of acute, active opportunistic infection, except oral thrush; oral, genital, or rectal herpes; and Mycobacterium avium bacteremia within 2 weeks prior to Screening Visit
* Currently have active malignant disease
* Significant ongoing or untreated abnormalities in cardiac, renal, hepatic, or pulmonary function that may interfere either with the ability to complete the study or the evaluation of adverse events
* Hypersensitivity to capsaicin (i.e., chili peppers or OTC capsaicin products), local anesthetics, Roxicodone®, Vicodin®, or adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-08; Study Completion 2005-11

PRIMARY OUTCOMES:
Percent change from baseline in the "average pain for the past 24 hours" Numeric Pain Rating Scale (NPRS) score (i.e., average of scores during Weeks 2-12, compared to baseline)

SECONDARY OUTCOMES:
Percent change from baseline in the "average pain for the past 24 hours" NPRS score (i.e., average of scores during Weeks 2-4 and 2-8, respectively, compared to baseline)
Proportion of subjects reaching 30% decrease from baseline in their "average pain for the past 24 hours" NPRS scores on average during Weeks 2-12, within each treatment group
Proportion of subjects reaching 30% decrease from baseline in their "average pain for the past 24 hours" NPRS scores on average during Weeks 2-4 and 2 8, respectively, within each treatment group
Percent change from baseline in the "worst pain for the past 24 hours" and "pain now" NPRS scores (baseline score compared to the average of scores from Weeks 2 -12), within each treatment group
"Pain now" on evening of treatment day
Mean onset and duration of efficacy in days within each treatment group
Proportion of subjects with significant changes in concomitant pain medication usage during Weeks 2-12, compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: David M Simpson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Jeffrey Tobias, MD, Study Director — NeurogesX
Locations (32):
- United States (32):
  - NeurogesX Investigational Site, Phoenix, Arizona
  - NeurogesX Investigational Site, Berkeley, California
  - NeurogesX Investigational Site, San Diego, California
  - NeurogesX Investigational Site, San Francisco, California
  - NeurogesX Investigational Site, Stanford, California
  - NeurogesX Investigational Site, West Hollywood, California
  - NeurogesX Investigational Site, Fort Lauderdale, Florida
  - NeurogesX Investigational Site, Miami, Florida
  - NeurogesX Investigational Site, North Palm Beach, Florida
  - NeurogesX Investigational Site, Orlando, Florida
  - NeurogesX Investigational Site, Sunrise, Florida
  - NeurogesX Investigational Site, Vero Beach, Florida
  - NeurogesX Investigational Site, Honolulu, Hawaii
  - NeurogesX Investigational Site, Chicago, Illinois
  - NeurogesX Investigational Site, Lexington, Kentucky
  - NeurogesX Investigational Site, Baltimore, Maryland
  - NeurogesX Investigational Site, Boston, Massachusetts
  - NeurogesX Investigational Site, Springfield, Massachusetts
  - NeurogesX Investigational Site, Detroit, Michigan
  - NeurogesX Investigational Site, Minneapolis, Minnesota
  - NeurogesX Investigational Site, St Louis, Missouri
  - NeurogesX Investigational Site, Camden, New Jersey
  - NeurogesX Investigational Site, Albany, New York
  - NeurogesX Investigational Site, New York, New York
  - NeurogesX Investigational Site, Chapel Hill, North Carolina
  - NeurogesX Investigational Site, Cleveland, Ohio
  - NeurogesX Investigational Site, Portland, Oregon
  - NeurogesX Investigational Site, Austin, Texas
  - NeurogesX Investigational Site, Dallas, Texas
  - NeurogesX Investigational Site, Houston, Texas
  - NeurogesX Investigational Site, San Antonio, Texas
  - NeurogesX Investigational Site, Madison, Wisconsin

REFERENCES:
- [Derived] Simpson DM, Brown S, Tobias JK, Vanhove GF; NGX-4010 C107 Study Group. NGX-4010, a capsaicin 8% dermal patch, for the treatment of painful HIV-associated distal sensory polyneuropathy: results of a 52-week open-label study. Clin J Pain. 2014 Feb;30(2):134-42. doi: 10.1097/AJP.0b013e318287a32f. PMID 23446088
- [Derived] Brown S, Simpson DM, Moyle G, Brew BJ, Schifitto G, Larbalestier N, Orkin C, Fisher M, Vanhove GF, Tobias JK. NGX-4010, a capsaicin 8% patch, for the treatment of painful HIV-associated distal sensory polyneuropathy: integrated analysis of two phase III, randomized, controlled trials. AIDS Res Ther. 2013 Jan 28;10(1):5. doi: 10.1186/1742-6405-10-5. PMID 23351618
- [Derived] Simpson DM, Brown S, Tobias J; NGX-4010 C107 Study Group. Controlled trial of high-concentration capsaicin patch for treatment of painful HIV neuropathy. Neurology. 2008 Jun 10;70(24):2305-13. doi: 10.1212/01.wnl.0000314647.35825.9c. PMID 18541884